CLINICAL TRIAL: NCT01221571
Title: A Pharmacodynamically-Guided Dose Escalation Phase I Study to Assess the Safety of AFM13 (Recombinant Antibody Construct Against Human CD30 and CD16A) in Patients With Refractory and/or Relapsed Hodgkin Lymphoma
Brief Title: A Study to Assess AFM13 in Patients With Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFM13-101; 2010-019232-13 (EudraCT Number)
Record Dates: First submitted 2010-10-05; First posted 2010-10-15 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2011-02

CONDITIONS: Hodgkin Lymphoma
Keywords: Phase I; Dose escalation; AFM 13; Natural killer cell
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFM13 (Experimental): IV (intravenous) infusion, dose escalation
  Interventions: Drug: AFM 13

INTERVENTIONS:
Drug: AFM 13 — Cohort escalation then expansion phase design. Starting dose 0.01 mg/kg. 4 weekly drug administrations.

SUMMARY:
The aim of this study is to determine the safety, tolerability, pharmacokinetics and activity of single cycles of AFM13 in patients with CD30 positive refractory and/or relapsed Hodgkin lymphoma.

DETAILED DESCRIPTION:
Study Objectives:

The overall objective of this study is to determine the safety, tolerability, pharmacokinetics and activity of single cycles of AFM13 in patients with CD30 positive refractory and/or relapsed Hodgkin lymphoma.

Objectives:

1. To determine the safety and tolerability of increasing doses of single cycles of AFM13 monotherapy.
2. To determine the OBD (Optimal Biological Dose) or MTD (Maximum Tolerated Dose) of AFM13; whichever is reached first.
3. To define the pharmacokinetic profile of AFM13.
4. To analyse immunological markers e.g. ADCC (Antibody dependent cell mediated cytotoxicity), NK (Natural killer) cell activity, complement activation and depletion, and cytokine release.
5. To assess the immunogenicity of AFM13.
6. To assess the activity of AFM13.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of relapsed or refractory Hodgkin lymphoma expressing the CD30 antigen.
2. Age ≥18 years.
3. Both genders.
4. Patients who have relapsed or are refractory after at least two prior potentially curative therapies including autologous stem cell transplantation (ASCT). Patients with a progressive disease after the first-line therapy who are ineligible for, or refused to receive high dose chemotherapy and/or ASCT for the second-line therapy, or any other established curative therapy, are also eligible.
5. Completed radiotherapy, chemotherapy, and/or treatment with other investigational agents at least 3 weeks prior to study entry.
6. Patients who received ASCT should have fully recovered prior to study entry.
7. Eastern Cooperative Oncology Group (ECOG) status of ≤2.
8. Laboratory data:

   1. Platelet count >75,000/mm3;
   2. Hemoglobin >9.0 g/dL (may be maintained by transfusion);
   3. Absolute neutrophil count >1500/mm3;
   4. ALT/AST (Alanine aminotransferase/Aspartate aminotransferase)<2.5 times the upper limit of normal (ULN);
   5. Total bilirubin <1.5 times ULN;
   6. Creatinine <1.5 mg/dL.
9. Female patients of childbearing potential who are not surgically sterile or postmenopausal and male patients who are not surgically sterile must agree to use medically effective contraception during the treatment period and up to 60 days after the last AFM13 administration. The patient must agree to sign his or her consent on this particular inclusion criterion.
10. Ability to give written, informed consent prior to any study-specific screening procedures, with the understanding that the consent may be withdrawn by the patient at any time without prejudice.
11. Be willing and able to comply with the study protocol for the duration of the study.

Exclusion Criteria:

1. Any significant diseases (other than HL (Hodgkin Lymphoma)) or clinically significant findings, including psychiatric and behavioral problems, medical history and/or physical examination findings that would preclude the patient from participating in the study.
2. History or clinical evidence of central nervous system (CNS) HL.
3. Allogeneic SCT.
4. Major surgery within 4 weeks prior to study entry.
5. Known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation.
6. Known history of another primary malignancy that has not been in remission for at least 5 years. Non-concurrent non-melanoma skin cancer and cervical carcinoma in situ or squamous intraepithelial lesions (e.g., cervical intraepithelial neoplasia [CIN] or prostatic intraepithelial/intraductal neoplasia [PIN]) are allowed.
7. Any active viral, bacterial, or systemic fungal infection within 4 weeks prior to study entry.
8. Known to be positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV).
9. History of significant chronic or recurrent infections requiring treatment.
10. Receiving systemic steroid prednisone or equivalent during the 3 weeks immediately preceding enrollment.
11. Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of AFM13 monotherapy. | Length of Study
  Measure occurrence of adverse events and monitor laboratory safety parameters. Immunogenicity of AFM13.

SECONDARY OUTCOMES:
To determine the OBD (Optimal Biological Dose) or MTD (Maximum Tolerated Dose) of AFM13 | Length of study
To define the pharmacokinetic profile of AFM13. | Length of study
  To test levels of AFM13 in blood samples and assess curve compared to dose of AFM13 administered.
To analyse immunological markers of activity | Length of study
  ADCC, NK cell, Complement and Cytokine levels in the serum will be measured at different time points to assess the level of activity resulting from administration of AFM13.
To assess the immunogenicity of AFM13. | length of study
To assess the activity of AFM13 | length of study
  To measure immunological activity useing biomarkers in the blood and to measure response of the disease in FDG-PET and CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Professor, Principal Investigator — University Hospital Cologne, Germany; Anas Younes, Professor, Principal Investigator — MD Anderson Cancer Center, Houston, Texas; Max S Topp, Professor, Principal Investigator — University Hospital Würzburg, Germany
Locations (3):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Germany (2):
  - University Hosptial Cologne, Cologne, Köln
  - University Hospital Würzburg, Würzburg

REFERENCES:
- [Derived] Rothe A, Sasse S, Topp MS, Eichenauer DA, Hummel H, Reiners KS, Dietlein M, Kuhnert G, Kessler J, Buerkle C, Ravic M, Knackmuss S, Marschner JP, Pogge von Strandmann E, Borchmann P, Engert A. A phase 1 study of the bispecific anti-CD30/CD16A antibody construct AFM13 in patients with relapsed or refractory Hodgkin lymphoma. Blood. 2015 Jun 25;125(26):4024-31. doi: 10.1182/blood-2014-12-614636. Epub 2015 Apr 17. PMID 25887777
- [Derived] Reiners KS, Kessler J, Sauer M, Rothe A, Hansen HP, Reusch U, Hucke C, Kohl U, Durkop H, Engert A, von Strandmann EP. Rescue of impaired NK cell activity in hodgkin lymphoma with bispecific antibodies in vitro and in patients. Mol Ther. 2013 Apr;21(4):895-903. doi: 10.1038/mt.2013.14. Epub 2013 Mar 5. PMID 23459515